CLINICAL TRIAL: NCT05941130
Title: Three-dimensional Evaluation of Postoperative Edema After Third Molar Surgery: a Randomized Clinical Trial
Brief Title: 3D Evaluation of Postoperative Edema After Third Molar Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: institutodeimplantologia
Record Dates: First submitted 2022-11-15; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Molar, Third; Third Molar Surgery; Soft Tissue Swelling; Pain, Postoperative; Quality of Life
Keywords: Third molar surgery; Three-dimensional imaging; postoperative Pain; Quality of Life; Oral surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutics; Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Patients assigned into group A (NSAID) will receive only Ibuprofen 600mg (Mylan)
  Interventions: Drug: Non-steroidal anti-inflammatory therapy (Ibuprofen 600mg Mylan)
- Group B (Experimental): Patients assigned into group B (CORT + NSAID) will receive Ibuprofen 600mg (Mylan) with methylprednisolone (Medrol, 16mg Pfizer Laboratories)
  Interventions: Drug: Combination of corticosteroid (methylprednisolone - Medrol, 16mg Pfizer Laboratories) therapy and non-steroidal anti-inflammatory (Ibuprofen 600mg Mylan) therapy

INTERVENTIONS:
Drug: Combination of corticosteroid (methylprednisolone - Medrol, 16mg Pfizer Laboratories) therapy and non-steroidal anti-inflammatory (Ibuprofen 600mg Mylan) therapy — Facial swelling assessment with a tridimensional method, pain and patient's quality of life will be evaluated after impacted third molar surgery, when NSAID are prescribed either alone (group A) or in combination with a corticosteroid (group B).Patients will be randomized before surgery into two groups regarding postoperative anti-inflammatory prescription.
  Half will receive postoperative steroid anti-inflammatory
  Other Names: CORT+NSAID
  Arms: Group B
Drug: Non-steroidal anti-inflammatory therapy (Ibuprofen 600mg Mylan) — Facial swelling assessment with a tridimensional method, pain and patient's quality of life will be evaluated after impacted third molar surgery, when NSAID are prescribed either alone (group A) or in combination with a corticosteroid (group B).Patients will be randomized before surgery into two groups regarding postoperative anti-inflammatory prescription.
  Half will receive postoperative non-steroid anti-inflammatory
  Other Names: NSAID
  Arms: Group A

SUMMARY:
Surgical removal of third molars is recognized as one of the most frequent procedures performed in oral surgery. Literature is rich in studies attempting to demonstrate the benefit of corticosteroids in third molar surgery, however the variety of methods, doses, routes and timing of administration has hampered the standardization of their use in light of best evidence. Also the use of 3D facial superimposition methodology to measure and analyze facial swelling after third molar surgery is a relatively new and promising technology.

DETAILED DESCRIPTION:
Surgical removal of third molars is recognized as one of the most frequent procedures performed in oral surgery. It is estimated that more than 50% of the population experience problems with their third molars, including impaction or other pathologies. Usually, recovery from third molar surgical procedures is straightforward, however some immediate side effects can be expected such as discomfort (pain), edema and trismus that are resolved within a few days. These results from postoperative tissue inflammatory response which present individual variations. Depending on the intensity of these postoperative symptoms and the severity of inflammatory response, daily activities may be temporarily affected and patient's overall quality of life might be impaired.

Factors as surgical technique, type of impaction, duration of the procedure, surgical complications and an inadequate pharmacotherapy may influence the severity of symptoms. Although edema and discomfort after the surgery cannot be completely eliminated, the possibility of reducing the frequency and severity of complications and improve patient's quality of life have been investigated.

Synthetic corticosteroids are widely used in surgery to control and reduce the post-surgical inflammatory response and pain since they limit inflammation and edema by reducing vascular dilatation and fluids transudation Literature is rich in studies attempting to demonstrate the benefit of corticosteroids in third molar surgery, however the variety of methods, doses, routes and timing of administration has hampered the standardization of their use in light of best evidence. To maximize the effectiveness in controlling both pain and swelling it is described in literature the combination of both NSAID and corticosteroids after third molar surgery, nevertheless reluctance and controversy regarding their coadministration in oral surgery still exists.

The use of 3D facial superimposition methodology to measure and analyze facial swelling after third molar surgery is a relatively new and promising technology that allows a high level of accuracy and a quantitative analysis of this outcome having a great potential to become the standard method for evaluating volumes and distances in facial and body anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals requiring surgical extraction of fully or partially impacted third molars requiring osteotomy;
* Individuals classified as grade I or II of the American Society of Anesthesiologists (ASA)
* Individuals with compliance to cooperate with the research protoco

Exclusion Criteria:

* Individuals with active bleeding or coagulation disorders
* Individuals with history of intolerance or hypersensitivity to the drugs included in the postoperative medication protocol
* Pregnant or lactating women
* Individuals with cysts or tumors around the embedded third molar
* Individuals who did not attend the control visits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Facial swelling | 7 postoperative days
  To evaluate postoperative facial swelling after impacted third molar surgery by using a 3D facial scanner in two different groups: A-NSAID alone; B - corticosteroid + NSAID. Each patient will perform three sets of facial soft tissue evaluation: before surgery (t0); 2 days postoperatively (t2) and 7 days postoperatively (t7). The changes in facial soft tissue volume after surgery will be qualitatively and volumetrically evaluated by using the previously validated 3D assessment with a 3D facial scanner (Bellus3D, version 2.2.1; Inc. Los Gatos, CA, USA) connected to a smartphone (Xiaomi Mi A2 Lite, Android version 9) via USB. Facial swelling will be determined by quantifying volumetric changes by using the superposition methodology and the alignment by the best fit algorithm of the pre and postoperative images, with Geomagic® software (Geomagic Inc., North Carolina, USA)

SECONDARY OUTCOMES:
Postoperative Pain | 7 postoperative days
  Postoperative pain will be assessed by using a Visual Analogue Scale (VAS) for pain. The Visual Analogue Scale for Pain ranges from 0 that represents "no pain" at the left pole to 100 (100mm scale) which represents 'worst imaginable pain" at the right pole Immediately before surgery, a form will be given to each patient with the scale and they will be instructed to place a line perpendicular to the Visual Analogue Scale line at the point that represents their level of pain at different times: immediately before surgery (t0), at review appointments on postoperative days 2 (t2) and 7 (t7).
  They will be also instructed to record the type and frequency of rescue medication taken to manage their pain levels.
Patient's quality of life | 7 postoperative days
  To assess oral health-related quality of life and to better understand patients' experience during the recovery period after third molar surgery, a short-form derivative of the Oral Health Impact Profile-49, the OHIP-14 will be used. The validated portuguese version of the selfreported 14-item Oral Health Impact Profile (OHIP-14) questionnaire will be completed by the patients before surgery (t0) and at postoperative days 2 (t2) and 7 (t7). The patients will be asked to respond according to frequency of impact on a 5-point Likert scale coded as: never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4) using a 12-months recall period.

CONTACTS AND LOCATIONS:
Overall Officials: João Caramês, DDS PhD, Study Director — Implantology Institute; Helena Francisco, DDS PhD, Study Chair — Implantology Institute; Catarina Pinto, DDS, Principal Investigator — Implantology Institute
Locations (1):
- Implantology Institute, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No